CLINICAL TRIAL: NCT02373293
Title: Epidemiologic , Observational, Prospective Study to Assess the Prognostic Value of the Antithrombin III in the Development of Moderate or Severe Acute Pancreatitis (AT-PROPANC)
Brief Title: Study to Assess the Prognostic Value of the Antithrombin III in the Acute Pancreatitis (AT-PROPANC)
Acronym: AT-PROPANC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Francisco Javier García Borobia (Other)
Collaborators: Alclinical Research, S.L. (Unknown)
Responsible Party: Sponsor-Investigator, Francisco Javier García Borobia, Dr., Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Other Study IDs: GAR-BOR/TAULI-2013
Record Dates: First submitted 2015-02-20; First posted 2015-02-27 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an epidemiological, observational, prospective, multicentric study in 400 adult patients admitted to hospital for mild acute pancreatitis to to assess the prognostic value of the antithrombin III in the development of moderate or severe acute pancreatitis.

DETAILED DESCRIPTION:
This is an epidemiological, observational, prospective, multicentric study in 400 adult patients admitted to hospital for mild acute pancreatitis to to assess the prognostic value of the antithrombin III in the development of moderate or severe acute pancreatitis.

In the context of clinical practice of general surgery and apparatus digestive services, patients entering with mild acute pancreatitis will be asked to participate in the study and if so, they will sign the informed consent.

On admission, demographic and anthropometric data of the patient will be recorded, as well as medical history, patient's admission data and vital signs. Patient's blood will be drawn for analysys and the risk of organ failure will be measured by modified Marshall and Apache II scales. The assessments and procedures performed are the standard practice at the center.

At 24 hours (± 3 hours) and at 7 days (or nine days to avoid weekends) after admisison, vital signs will be recorded, laboratory tests will be performed and the risk of organ failure will be measured by modified Marshall and Apache II scales.

At discharge of the patient (regardless of when it occurs), the outcome of the acute pancreatitis will be recorded.

. Those patients discharged within the first month after admission will be visited or called (according to standard practice at the center) one month after arrival, to record follow-up data, including health condition, readmissions and abdominal pain evaluation by visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild acute pancreatitis according to seriousness criteria established by Banks et al, 2013.
* Patients of either sex aged ≥ 18 years .
* Patients who have given their written informed consent

Exclusion Criteria:

* Patients with exacerbated chronic pancreatitis.
* Patients with coagulation disorders (congenital and acquired antithrombin deficiency) .
* Patients with liver cirrhosis.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with mild acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-01-18; Primary Completion 2015-01-30 (Actual); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
antithrombin III levels vs maximum seriousness grade of acute pancreatitis | At Admission and at 24h
  Levels of antithrombin III at admission and at 24h will be related with maximum seriousness grade of acute pancreatitis reached during patient's admission at site by logistic regression models

SECONDARY OUTCOMES:
result of modified Marshall and Apache II scales | Admission and at 24h
antithrombin III levels vs mortality | From date of admission until the end of study or date of death from any cause, whichever came first, assessed up to 1 month"
  Levels of antithrombin III at admission and at 24h will be related with mortality rates by logistic regression models
antithrombin III levels vs organic failure | From date of admission until the end of study or date of organic failure, whichever came first, assessed up to 1 month"
  Levels of antithrombin III at admission and at 24h will be related with organic failure rates by logistic regression models
antithrombin III levels vs necrosis and infection rates | From date of admission until the end of study or date of necrosis or infection diagnosis, whichever came first, assessed up to 1 month"
  Levels of antithrombin III at admission and at 24h will be related with necrosis and infection rates by logistic regression models

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier García Borobia, Dr., Principal Investigator — Corporacion Parc Tauli
Locations (2):
- Spain (2):
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital de Sant Joan Despí Moisés Broggi, Sant Joan Despí, Barcelona

REFERENCES:
- [Derived] Garcia Borobia F, Flores Clotet R, Bejarano Gonzalez N, Gonzalez Martinez S, Garcia Monforte N, Romaguera Monzonis A, Gonzalez Abos C, Gonzalez Abos S, Lucas Guerrero V, Perez Perarnau A, Mota Villaplana F. Predictive Value of Antithrombin III and d -Dimer in the Development of Moderate-To-Severe Acute Pancreatitis : A Prospective, Observational Study (AT-PROPANC). Pancreas. 2023 Apr 1;52(4):e241-e248. doi: 10.1097/MPA.0000000000002245. Epub 2023 Sep 20. PMID 37801622